CLINICAL TRIAL: NCT06742203
Title: WPMDE1 - Whey Protein Milk-Derived Exosomes Among Healthy Subjects- a Phase 1, Single-center, Open-label Study
Brief Title: WPMDE1 - Whey Protein Milk-Derived Exosomes Among Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Exosomm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WPMDE1
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: IBD

STUDY DESIGN:
Intervention Model Description: Tolerability: Identification of dose ranges that do not cause discomfort or adverse symptoms over the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exosomm treatment (Experimental): Experimental Group: WPMDE1 - Whey Protein Milk-Derived Exosomes
  Administered as a powder dissolved in water and taken orally twice daily in pre-measured sachets.
  Interventions: Dietary Supplement: Whey Protein Milk-Derived EVs

INTERVENTIONS:
Dietary Supplement: Whey Protein Milk-Derived EVs — WPMDE1 - Whey Protein Milk-Derived EVs, is a white powder obtained by filtration, concentration, and dehydrating whey solution, with the addition of sweeteners and flavorings to balance the taste. The WPMDE1 contains a known concentration of EVs (also known as milk exosomes).

SUMMARY:
This phase 1, single-center, open-label study aims to evaluate the tolerability and usability of WPMDE1, a whey protein milk-derived exosome (EV) nutritional supplement, in healthy adults. The study will assess dose tolerability and determine the appropriate dosage for future studies targeting patients with Irritable Bowel Syndrome (IBS) and Inflammatory Bowel Disease (IBD).

DETAILED DESCRIPTION:
WPMDE1 is a nutritional supplement derived from cow's milk using a novel production process designed to preserve extracellular vesicles (EVs) and their biological functions. This single-arm, unblinded trial will explore the effects of ascending doses of WPMDE1 on tolerability and usability in up to 30 healthy adults aged 18-60. Participants will be divided into five groups to test incremental doses over 7-30 days.

The study includes blood sampling, vital sign measurements, and daily symptom tracking via validated gastrointestinal symptom questionnaires. The outcomes will inform the design of future clinical trials targeting IBS and IBD patients. The trial will be conducted at Hadassah University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants who have not undergone any major surgeries or hospitalization 6 months prior to entering the study
* All genders
* Participants aged 18-60
* Participants with no underlying known health or mental conditions
* Participants who are not participating in another clinical study simultaneously or taking any other nutritional supplements or chronic drugs.
* Participants must pre-sign the informed consent form.

Exclusion Criteria:

* Participants who violate one or more of the inclusion criteria
* participants with chronic diseases, particularly those that are related to the GI tract
* Participants with cow milk allergy/ intolerance or history of such.
* Participants suffering from constipation or diarrhea
* Participants who use drugs or drink alcohol on a regular basis (more than one glass per week)
* Pregnant or breastfeeding women
* Participants with a BMI over 30

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Tolerability of adverse symptoms over the study period. | up to 30 days
  Tolerability: Identification of dose ranges that do not cause discomfort or adverse symptoms over the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel